CLINICAL TRIAL: NCT05788783
Title: Evaluating the Impact of a Canine-assisted Therapy Program in Youth Enrolled in Outpatient Treatment for Social, Emotional, and Behavioral Problems.
Brief Title: Feasibility of a Dog Training Therapy Program in UC Outpatient Youth Receiving Psychiatric Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Canine-Therapy Corp (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB22-1218
Record Dates: First submitted 2023-01-30; First posted 2023-03-29 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-03

CONDITIONS: Emotion Regulation; Behavioral Disorder; Self Esteem
MeSH Terms: conditions — Emotional Regulation; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Active intervention. Youth will be assigned to the active Recovery & Care Canine-Assisted Therapy intervention arm.
  Interventions: Behavioral: Recovery & Care Canine-Assisted Therapy
- Active control (Other): Active control intervention. Youth will be assigned to the active Canine Education & Bonding arm.
  Interventions: Other: Canine Education & Bonding

INTERVENTIONS:
Behavioral: Recovery & Care Canine-Assisted Therapy — Active intervention. An 6-week session of structured, goal-oriented activities where youth focus on mastering dog obedience and dog training skills. Each session is 1 hour and 15 minutes in length and includes education, review of prior sessions, and specific skill-building activities. Skill-building activities progress in complexity during the course of the 6-week curriculum.
  Arms: Experimental
Other: Canine Education & Bonding — Active control intervention. An 6-week session of semi-structured activities. Sessions are 45 minutes in length. Youth in this condition engage in an educational component, passive observation of dog-training skills, and an active free-play session with the dog-handler teams.
  Arms: Active control

SUMMARY:
The goal of this pilot project is to test for initial efficacy of the Recovery & Care Canine-Assisted Therapy program that has been developed and implemented in Lawrence Hall, a Chicago-based residential treatment center for maltreated youth. In this study, the investigators test the feasibility, acceptability, and short-term efficacy of expanding the program to a group of youth currently in outpatient treatment for social, emotional, and behavioral problems. Results from this project will provide preliminary evidence of whether a structured, goal-oriented intervention program focused on dog training activities has direct impact on increasing youth emotional self-regulation, impulse control, and self-efficacy, which are important targets for intervention among youth with mental health problems. If successful, this project could lead to a larger, randomized control clinical trials study that tests the longitudinal impact of the program that could further lead to national dissemination of the Recovery & Care curriculum as an alternative therapeutic approach.

DETAILED DESCRIPTION:
The study uses a longitudinal, within-person design with two parallel conditions. This study involves three cohorts of youth who will participate in one of two 6-week interventions. For each cohort of youth, half of the sample will be randomly assigned to the Recovery & Care Canine-Assisted Therapy condition, and half of the sample will be randomly assigned to an active control condition (Canine Education & Bonding). The two conditions will run in parallel. The order of the two intervention conditions will be counterbalanced across study cohorts.

The Recovery & Care Canine-Assisted Therapy intervention is a 1.25 hour structured curriculum that will occur weekly across a period of 6 weeks. The program will be delivered by the Canine Therapy Corps (CTCorps) offsite at the CtCorps facility. Youth will work with CTC-affiliate staff, including trained dog-handler teams, a canine behavior expert, and a clinical supervisor to engage in a series of structured activities progress throughout the intervention. Week 1 is a "meet-and-greet" session where youth are introduced to all dog-handler teams participating in the program and will be asked to select a team to work with for the following sessions. Each youth is assigned their own dog-handler team. Weeks 2 cover activities regarding dog obedience, building from mastering basic commands which the dog already knows (such as "sit," "stay'") to the introduction of "new tricks" that the dog has not yet learned. In Weeks 3, youth will continue to work on mastering the "new tricks" with their dog-handler team and will also begin dog agility training. The agility training session progress in terms of complexity of number and types of obstacles. Week 4 is for proofing all skills (obedience, trick, agility) learned in previous sessions. Week 5 continues proofing all skills and is discussion of the graduation structure and dress rehearsal, and Week 6 is a graduation ceremony where family and friends are invited to observe the progress each youth has made with their dog-handler team. In Weeks 1-5, the goals of each session are outlined at the beginning of the session and brief education is provided regarding the session goals. Weeks 2-5 also include a review of the skills/activities covered in prior weeks. At the end of sessions 1-5, youth are asked to reflect on what they did during the session, including discussion of what they did really well, what they wanted to work on further, and goals for the next session. Research staff will be present during all sessions to record fidelity measures. The Positive and Negative Affect Scale will be administered on-site by research staff at the beginning and end of each intervention session. Change in affect are primary and secondary outcome measures.

The Canine Education & Bonding intervention is a series of 45-minute, semi-structured activities that will occur weekly across the same 6-week period as the Recovery & Care intervention. Youth will work with the same group of CTCorps-affiliate staff involved the Recovery & Care intervention, including the same set of dog-handler teams. These sessions will begin with education on basic aspects of dogs (e.g., different breed types, caring for dogs, etc.). Youth will then passively observe the dog-handler teams demonstrating basics of dog obedience and dog agility training that parallel that activities done in the Recovery & Care Canine-Assisted Therapy session that same week. Following the education and passive demonstration sessions, youth will be allowed to interact freely with the dog-handler teams. A brief mood questionnaire will be administered by research staff at the beginning and end of each session. Research staff will also be present during all sessions as observers and to record fidelity measures.

Baseline and Follow-up data will be collected up to 1-month before and 1-month after the intervention programs. Data collection for all subjects enrolled will be conducted by the University of Chicago Project staff, on site in the PI's lab at the University of Chicago or virtually.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving outpatient mental health services at the University of Chicago or have received outpatient mental health services from the community in the last 12 months.
* Available for scheduling during the entire 6-week intervention program
* Interest in participating in the program

Exclusion Criteria:

* Severe cognitive, psychiatric, or physical condition or limitation that would prevent participation.
* Severe animal allergy
* Animal phobia
* History of mistreatment of animals.
* Above-average scores on both measures of behavioral regulation and emotional regulation
* WASI t-score of intellectual ability < 60.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Emotional Stroop | Up to 1-month post-intervention
  Computer-Assisted task assessing affect regulation
Change in Emotional Stroop | Change from baseline to up to 1-month post-intervention
  Computer-Assisted task assessing affect regulation
Flanker Task | Up to 1-month post-intervention
  Computer-Assisted task assessing attention & inhibitory control
Change in Flanker Task | Change from baseline to up to 1-month post-intervention
  Computer-Assisted task assessing attention & inhibitory control
Rosenberg Self-Esteem Scale | Up to 1-month post-intervention
  10-item self-report scale assessing self-esteem. Higher scores are better outcomes
Change in Rosenberg Self-Esteem Scale | Change from baseline to up to 1-month post-intervention
  10-item self-report scale assessing self-esteem. Higher scores are better outcomes
Change in Negative Affect | Change from the beginning to the end of each of the 6 weekly intervention sessions
  In addition to overall change in outcomes post intervention, we are also interested in whether each intervention session produces an immediate change in youth emotion. We will assess negative affect using 5 self-report items on current mood from positive and negative affect scale. Higher scores are worse outcomes.

SECONDARY OUTCOMES:
Pearson Social Skills Rating Scales -Positive social behaviors | Up to 1-month post-intervention
  Self-report subscale assessing cooperation, empathy, assertion, self-control, and responsibility. Higher scores are better outcomes.
Change in Pearson Social Skills Rating Scales -Positive social behaviors | Change from baseline to up to 1-month post-intervention
  Self-report subscale assessing cooperation, empathy, assertion, self-control, and responsibility. Higher scores are better outcomes.
Pearson Social Skills Rating Scales -Externalizing behaviors | Up to 1-month post-intervention
  Self-report subscale assessing aggressive acts and poor temper control. Higher scores are worse outcomes
Change in Pearson Social Skills Rating Scales -Externalizing behaviors | Change from baseline to up to 1-month post-intervention
  Self-report subscale assessing aggressive acts and poor temper control. Higher scores are worse outcomes
Attendance and Attrition | Aggregated across the 6-week intervention program
  Project staff will record the number of absences and drop-outs for youth enrolled in both study intervention conditions.
Change in Positive Affect | Change from the beginning to the end of each of the 6 weekly intervention session
  In addition to overall change in outcomes post intervention, we are also interested in whether each intervention session produces an immediate change in youth emotion. We will assess positive affect using 5 self-report items on current mood from positive and negative affect scale. Higher scores are better outcomes.
Self-Regulation Child Report | Up to 1-month post-intervention
  Behavioral and emotional regulation subscales from the BRIEF-2 instrument
Self-Regulation Parent Report | Up to 1-month post-intervention
  Behavioral and emotional regulation subscales from the BRIEF-2 instrument

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05788783/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT05788783/ICF_001.pdf